CLINICAL TRIAL: NCT02750410
Title: A Phase 4 Study of Efficacy and Safety of Dulaglutide When Added to Insulin Treatment With or Without Oral Antidiabetic Medication in Patients With Type 2 Diabetes
Brief Title: A Study of Dulaglutide in Japanese Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15803; H9X-JE-GBGF (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dulaglutide (Experimental): Dulaglutide 0.75 milligram (mg) administered once weekly for 16 weeks. After 16-weeks, dulaglutide administered once weekly for 36 weeks.
  Interventions: Drug: Dulaglutide
- Placebo (Placebo Comparator): Placebo administered once weekly for 16 weeks. After 16-weeks, dulaglutide 0.75 mg administered once weekly for 36 weeks.
  Interventions: Drug: Dulaglutide; Drug: Placebo

INTERVENTIONS:
Drug: Dulaglutide — Administered subcutaneously (SC)
  Other Names: LY2189265
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of combination therapy with dulaglutide and insulin in Japanese participants with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have had a diagnosis of type 2 diabetes mellitus
* Participants who have been treated with insulin therapy (basal insulin, premixed insulin, or basal/mealtime insulin regimen) with or without 1 or 2 oral antidiabetics (OADs) at stable dose for at least 3 months before screening
* Participants who have an HbA1c value ≥7.0% and ≤10.5% at screening if the participant is washing out OADs (dipeptidyl peptidase-4 [DPP-4] inhibitors, sulfonylurea [SU], or glinides) or ≥7.5% and ≤10.5% at screening if the participant is not washing out OADs
* Participants who have stable weight (±5%) ≥3 months prior to screening
* Participants who have a body mass index (BMI) of 18.5 to 35.0 kilograms per meter squared (kg/m^2)

Exclusion Criteria:

* Participants who have a diagnosis of type 1 diabetes
* Participants who have previously received therapy with a glucagon-like peptide-1 receptor agonist within 3 months prior to screening
* Participants who have been previously treated with dulaglutide prior to screening
* Participants who have been treated with 2 of the following at screening: DPP-4 inhibitor, SU, and glinide (ie, DPP-4 inhibitor and SU, or DPP-4 inhibitor and glinide)
* Participants who have been treated with continuous subcutaneous insulin infusion (CSII) at screening
* Participants who have clinically significant gastric emptying abnormality, hepatitis, pancreatitis, renal dysfunction, or thyroid abnormalities
* Participants who have a history of clinically significant cardiovascular disease, transplanted organ, or active or untreated malignancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-08; Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- Japan (25):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adachi-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiyoda City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chuou-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chūōku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chūōku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fuchū
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ichikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Isahaya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kamakura
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kashihara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maebashi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Mito
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Naka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nishinomiya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sasebo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Shimotsuke
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Onishi Y, Ishii H, Oura T, Takeuchi M. Efficacy and Safety of Once-Weekly Dulaglutide in Type 2 Diabetes Patients Using Insulin: Exploratory Subgroup Analysis by Insulin Regimen. Diabetes Ther. 2020 Mar;11(3):735-745. doi: 10.1007/s13300-020-00765-6. Epub 2020 Jan 29. PMID 31994009
- [Derived] Ishii H, Onishi Y, Oura T, Takeuchi M. Once-Weekly Dulaglutide with Insulin Therapy for Type 2 Diabetes: Efficacy and Safety Results from a Phase 4, Randomized, Placebo-Controlled Study. Diabetes Ther. 2020 Jan;11(1):133-145. doi: 10.1007/s13300-019-00726-8. Epub 2019 Nov 22. PMID 31758520

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After 16 weeks of the primary double-blind treatment period, participants taking placebo were switched to dulaglutide for an additional 36 weeks of open-label extension treatment. Efficacy was assessed for 16 weeks based on hypoglycemic agent evaluation.
Groups:
- Placebo: Placebo administered subcutaneously (SC) once weekly for 16 weeks. After 16-weeks, Dulaglutide 0.75 milligram (mg) administered SC once weekly for 36 weeks.
- Dulaglutide: Dulaglutide administered SC once weekly for 16 weeks. After 16-weeks, Dulaglutide 0.75 mg administered SC once weekly for 36 weeks.
Period: Double-Blind Treatment Period
Arm/Group | Placebo | Dulaglutide
Started | 39 | 120
Received at Least One Dose of Study Drug | 39 | 120
Completed | 37 | 117
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Open-Label Extension Period
Arm/Group | Placebo | Dulaglutide
Started | 37 | 117
Completed | 31 | 111
Not Completed | 6 | 6
Not completed — Adverse Event | 5 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Placebo administered SC once weekly for 16 weeks. After 16-weeks, Dulaglutide 0.75 mg administered SC once weekly for 36 weeks.
- Dulaglutide: Dulaglutide 0.75 mg administered SC once weekly for 16 weeks. After 16-weeks, Dulaglutide 0.75 mg administered SC once weekly for 36 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dulaglutide | Total
Number analyzed (Participants) | 39 | 120 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.68) | 59.3 (10.23) | 59.3 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 42 | 61
  Male | 20 | 78 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 120 | 159
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 39 | 120 | 159
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 39 | 120 | 159
Percentage of Hemoglobin A1c (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.64 (0.72) | 8.50 (0.69) | 8.53 (0.70)
Percentage of Participants with Insulin regimen [Number; unit: percentage of insulin regimen]
  Basal | 43.6 | 43.3 | 43.4
  Premixed | 23.1 | 21.7 | 22.0
  Basal/meal time | 33.3 | 35.0 | 34.6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least square (LS) mean in HbA1c was calculated using a restricted maximum likelihood (REML) based mixed-effects model for repeated measures (MMRM) and adjusted by, baseline HbA1c, treatment, visit, and treatment-by-visit insulin regimen (basal insulin, premixed insulin, or basal/mealtime insulin), where participant treated as a random effect.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline HbA1c.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Placebo: Placebo administered SC for 16 weeks.
- Dulaglutide: Dulaglutide 0.75 mg administered SC once weekly for 16 weeks.
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 39 | 120
percentage of HbA1c | 0.06 (0.099) | -1.45 (0.057)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean percent difference = -1.50, 95% CI 2-sided [-1.73 to -1.28]

2. Secondary Outcome: Percentage of Participants With HbA1c <7.0% or ≤6.5%
Description: Percentage of participants whose HbA1c was <7.0% or ≤6.5%. HbA1c <7.0% is presented.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug had evaluable post-baseline HbA1c data. HbA1c ≤6.5% had no results since model did not converge.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 36 | 116
percentage of participants | 47.4 | 0
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; analysis was based on repeated measures logistic regression; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 0.117, 95% CI 2-sided [0.028 to 0.479]

3. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG)
Description: The LS mean change from baseline in FSG was calculated using a REML based MMRM and adjusted by, baseline value, treatment, visit, treatment-by-visit, baseline HbA1c Group (<8.5%, >=8.5%) + insulin regimen (basal insulin, premixed insulin, or basal/mealtime insulin), where participant treated as a random effect.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had evaluable post baseline data.
Measure: Least Squares Mean (Standard Error); unit: milligram/deciliter (mg/dL)
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 39 | 118
milligram/deciliter (mg/dL) | -4.1 (4.94) | -34.2 (2.78)
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -30.14, 95% CI 2-sided [-41.37 to -18.91]

4. Secondary Outcome: Change From Baseline in Plasma Glucose From 7-Point Self-Monitored Blood Glucose Profiles (SMBG)
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: prebreakfast blood glucose (BG), breakfast 2-hour postprandial blood glucose (PPBG), prelunch BG, lunch 2-hour PPBG, predinner BG, dinner 2-hour PPBG, and bedtime BG. LS mean was calculated with fixed effect test of analysis of covariance (ANCOVA) model and adjusted by, baseline value, treatment, baseline HbA1c Group (<8.5%, ≥8.5%), insulin regimen (basal insulin, premixed insulin, or basal/mealtime insulin).
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had evaluable post baseline data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Placebo; Dulaglutide: Placebo administered SC once weekly for 16 weeks.
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 39 | 120
mg/dL
  Prebreakfast BG: number analyzed (Participants) | 37 | 115
  Prebreakfast BG | 12.30 (4.37) | -14.28 (2.52)
  Breakfast 2-hour PPBG: number analyzed (Participants) | 36 | 114
  Breakfast 2-hour PPBG | 13.15 (7.35) | -32.24 (4.19)
  Prelunch BG: number analyzed (Participants) | 36 | 114
  Prelunch BG | 8.08 (5.56) | -28.74 (3.18)
  Lunch 2-hour PPBG: number analyzed (Participants) | 36 | 114
  Lunch 2-hour PPBG | 10.74 (7.39) | -39.42 (4.54)
  Predinner BG: number analyzed (Participants) | 36 | 115
  Predinner BG | 5.66 (5.74) | -25.61 (3.28)
  Dinner 2-hour PPBG: number analyzed (Participants) | 36 | 116
  Dinner 2-hour PPBG | 3.97 (7.91) | -30.99 (4.48)
  Bedtime BG: number analyzed (Participants) | 34 | 107
  Bedtime BG | 13.21 (7.78) | -28.24 (4.45)
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; Prebreakfast BG; Test type: Superiority; p < 0.001, t-test, 2 sided; LS mean difference = -26.59, 95% CI 2-sided [-36.39 to -16.78]
Statistical Analysis 2: Comparison: Placebo vs Dulaglutide; Breakfast 2-hour PPBG; Test type: Superiority; p < 0.001, t-test, 2 sided; LS mean difference = -45.38, 95% CI 2-sided [-61.77 to -29.00]
Statistical Analysis 3: Comparison: Placebo vs Dulaglutide; Prelunch BG; Test type: Superiority; p < 0.001, t-test, 2 sided; LS mean difference = -36.82, 95% CI 2-sided [-49.20 to -24.45]
Statistical Analysis 4: Comparison: Placebo vs Dulaglutide; Lunch 2-hour PPBG; Test type: Superiority; p < 0.001, t-test, 2 sided; LS mean difference = -50.16, 95% CI 2-sided [-67.85 to -32.46]
Statistical Analysis 5: Comparison: Placebo vs Dulaglutide; Predinner BG; Test type: Superiority; p < 0.001, t-test, 2 sided; LS mean difference = -31.27, 95% CI 2-sided [-44.05 to -18.48]
Statistical Analysis 6: Comparison: Placebo vs Dulaglutide; Dinner 2-hour PPBG; Test type: Superiority; p < 0.001, t-test, 2 sided; LS mean difference = -34.97, 95% CI 2-sided [-52.55 to -17.38]
Statistical Analysis 7: Comparison: Placebo vs Dulaglutide; Bedtime BG; Test type: Superiority; p < 0.001, t-test, 2 sided; LS mean difference = -41.45, 95% CI 2-sided [-58.81 to -24.09]

5. Secondary Outcome: Change From Baseline in Body Weight
Description: LS mean change from baseline in body weight was calculated using a REML based MMRM and was adjusted by, baseline value, treatment, visit, treatment-by-visit, baseline HbA1c group (<8.5%, >=8.5%), insulin regimen (basal insulin, premixed insulin, or basal/mealtime insulin), where participant treated as a random effect.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had evaluable post baseline data.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 39 | 120
kilogram (kg) | -0.30 (0.302) | -0.20 (0.171)
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; Test type: Superiority; p = 0.776, Mixed Models Analysis; LS mean difference = 0.10, 95% CI 2-sided [-0.59 to 0.78]

6. Secondary Outcome: Change From Baseline in Daily Total Insulin Dose
Description: Mean change from baseline in total insulin dose was measured in each treatment groups.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: International Units (IU)/Day
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 39 | 120
International Units (IU)/Day | -0.3 (1.2) | -1.1 (3.1)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: All randomized participants who received at least one dose of study drug in the double-blind treatment period and continued to open-label extension period.
Groups:
- Placebo Double-Blind (DB) Treatment Period: Placebo administered SC once weekly for 16 weeks.
- Dulaglutide 0.75 mg DB Treatment Period: Dulaglutide 0.75 mg administered SC once weekly for 16 weeks.
- Placebo DB Treatment, Dulaglutide 0.75 mg Extension Period: Placebo administered SC once weekly for 16 weeks then Dulaglutide 0.75 mg administered SC once weekly for 36 weeks.
- Dulaglutide 0.75 mg DB Treatment/Extension Period: Dulaglutide 0.75 mg administered SC once weekly for 52 weeks.
Arm/Group | Placebo Double-Blind (DB) Treatment Period | Dulaglutide 0.75 mg DB Treatment Period | Placebo DB Treatment, Dulaglutide 0.75 mg Extension Period | Dulaglutide 0.75 mg DB Treatment/Extension Period
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/120 | 0/39 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/39 | 3/120 | 1/39 | 6/120
Other Adverse Events (participants affected / at risk) | 18/39 | 47/120 | 28/39 | 59/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double-Blind (DB) Treatment Period (N=39) | Dulaglutide 0.75 mg DB Treatment Period (N=120) | Placebo DB Treatment, Dulaglutide 0.75 mg Extension Period (N=39) | Dulaglutide 0.75 mg DB Treatment/Extension Period (N=120)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double-Blind (DB) Treatment Period (N=39) | Dulaglutide 0.75 mg DB Treatment Period (N=120) | Placebo DB Treatment, Dulaglutide 0.75 mg Extension Period (N=39) | Dulaglutide 0.75 mg DB Treatment/Extension Period (N=120)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 10 (17) | 5 (5) | 11 (18)
Constipation (Gastrointestinal disorders) | 4 (4) | 8 (8) | 5 (5) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (6) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (8) | 2 (2) | 7 (8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 3 (3) | 6 (7)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 5 (6)
Nasopharyngitis (Infections and infestations) | 7 (8) | 19 (22) | 12 (15) | 34 (49)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (3) | 2 (2) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 8 (8) | 2 (2) | 9 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT02750410/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT02750410/SAP_001.pdf